CLINICAL TRIAL: NCT00722280
Title: The Pittsburgh Protocol in Human Upper Extremity Allotransplantation
Brief Title: Human Upper Extremity (Hand and Forearm) Allotransplantation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: loss of funding
Sponsor: University of Pittsburgh (Other)
Collaborators: Armed Forces Institute of Regenerative Medicine (U.S. Federal Agency); U.S. Army Medical Research and Development Command (U.S. Federal Agency); San Antonio Military Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Mario Solari, Assistant Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO07030180
Record Dates: First submitted 2008-07-23; First posted 2008-07-25 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Amputation, Traumatic
Keywords: Amputation, upper limb, composite tissue, immunosuppression
MeSH Terms: conditions — Amputation, Traumatic | interventions — Hand Transplantation; Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hand Transplantation (Experimental): Described above
  Interventions: Procedure: Hand Transplantation

INTERVENTIONS:
Procedure: Hand Transplantation — This program is the primary site for a novel immune modulation protocol for hand and/or forearm transplantation using donor bone marrow stem cells. This protocol, otherwise called the "Pittsburgh Protocol" has been published and implemented in 8 hand/forearm transplantations. The Pittsburgh hand transplant program is the only center that has experience with the "Pittsburgh Protocol" to reduce the number and dosing of immunosuppressive drugs used to prevent rejection of hand/forearm transplants.
  Other Names: Induction Immunosuppression; Maintenance Immunosuppression; Surgical Transplantation of Human Hand or Forearm; Rehabilitation

SUMMARY:
Overall Goal

To establish hand transplantation as a safe and effective reconstructive strategy for the treatment of upper extremity amputations.

Specific Aim

To reduce the risk of rejection and enable allograft survival while minimizing the requirement for long term high dose immunosuppression.

For this purpose, we propose to utilize the "Pittsburgh Protocol", which is an immunomodulatory strategy that has been implemented in solid organ transplants at UPMC. Early results in living related liver and kidney patients have confirmed that this protocol provides the means to allow graft survival with minimization of maintenance immunosuppression and even allows weaning of some patients from long-term immunosuppression.We hypothesize that a similar protocol can enable graft survival in highly immunogenic composite tissue allografts like hand transplants while reducing the number,dosing and/or frequency of immunosuppressive drugs associated with serious adverse effects.

DETAILED DESCRIPTION:
Suitable candidates will be identified via patient information brochures and via advertisements directed at upper limb amputees. For this purpose, a web-page will be constructed for free access by interested individuals. This website will be accessible through standard search engines. Interested potential subjects will be instructed to contact the investigator for an appointment. At the time of appointment, candidates will be first requested to complete a screening consent form (SCF) before undergoing further evaluation/medical screening procedures. The SCF includes a written consent to obtain PHI of the candidate. When the candidate visits UPMC he will undergo a consultation with the PI who will perform a thorough clinical assessment and explain in detail the treatment options, risks and benefits of the procedure. Candidates will be requested to complete a screening consent at this stage. Appropriate subjects will then undergo further medical screening procedures that include a number of examinations and investigations to determine their candidacy for hand transplantation. Prospective recipients who are selected based on results of screening procedures will be invited to review and sign the full informed consent form prior to being wait-listed for the procedure.

The screening tests include:

History and physical exam, including height and weight Urine pregnancy test for all female subjects of childbearing potential Complete blood count, differential, reticulocyte count, platelet count ABO type Liver function tests including SGPT or SGOT, serum bilirubin (total and direct), total protein, albumin, alkaline phosphatase and GGT, PT, PTT with INR Serum electrolytes and renal function panel to include the following: sodium, potassium, chloride, carbon dioxide, calcium, phosphorus, magnesium, glucose, creatinine and BUN Urinalysis and creatinine clearance test to determine GFR Infectious disease studies: HIV antigen, HTLV I-II antibody, antibodies to HIV 1 and 2, hepatitis C virus, syphilis, hepatitis B core antibody, and hepatitis B surface antigen titers are required Infectious disease titers: CMV, EBV, HSV, toxoplasmosis and VZV (IgG and IgM when indicated) Pulmonary function tests, including DLCO2 Chest X-ray EKG and MUGA scan or echocardiogram for determination of cardiac ejection fraction Sinus X-ray (if clinically indicated) CT scans (CT Angiography)/MRI studies (Functional MRI, Skeletal MRIs of hand/hips) as indicated by medical history and physical examination Ophthalmologic examination Dental consult Psychiatric evaluation

ELIGIBILITY:
Donor Selection Criteria

Brain dead donors who have met the criteria for Determination of Death will be selected by the hand transplant team in conjunction with the CORE (Center for Organ Recovery and Education), the organ procurement agency (OPO) for Pittsburgh and covers Pennsylvania, New York and West Virginia. The mandatory requirements are family consent for limb donation, stable donor (does not require excessive vasopressors to maintain blood pressure), age between 18 to 55 years, limb matched for size with recipient, same blood type as recipient, negative cross-match, and importantly accurately matched for gender, skin tone and race (may be relative requirement depending on recipient consent).

Recipient Selection Criteria

Recipients will be selected from a population of subjects with upper limb loss. Recipients may be male or female and of any race, color or ethnicity.

Inclusion Criteria:

1. Age (>18 years <60 years): Recipients <18 years of age are excluded due to limitations of giving full informed consent and the potentially increased risk of lymphoproliferative disorder in a younger population. Once hand transplantation and in particular the strategy for minimizing immunosuppression has proven to be efficacious and safe, the restrictions with regard to recipient age may be relaxed.
2. No serious co-existing medical (coronary artery disease, diabetes) or psycho-social problems (including alcoholism, drug abuse).
3. Must be negative for malignancy (for 10 years) or HIV (at transplant).
4. Negative crossmatch with donor.
5. Negative pregnancy test in female recipient of child bearing potential and consent to use reliable contraception for at least one year following transplantation.
6. Consent to cell collection, storage, and bone marrow infusion as part of the treatment regime.
7. Amputation may be recent (acute injury) or remote (patient may have undergone rehabilitation with prostheses).

Exclusion Criteria:

1. Conditions that may impact the immunomodulatory protocol: These include diseases like HIV or malignancy that could expose the recipient to an unacceptable risk under immunosuppressive treatment. Sensitized recipients with high level of preformed antibodies are also at risk.
2. Conditions that may impact the success of the surgical procedure or increase the risk of postoperative complications: These include inherited coagulopathies like Hemophilia, Von-Willebrand's disease, Protein C and S deficiency, Thrombocythemias, Thallassemias, Sickle Cell disease etc. Mixed connective tissue diseases and collagen diseases can result in poor wound healing after surgery,
3. Conditions that may impact functional outcomes: Lipopolysaccharidoses and amyloidosis are few of the conditions that may impact nerve regeneration and impair outcomes. Also, rare disorders of bone healing like osteopetrosis may also be causes for exclusion.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2008-12; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Graft survival | One to ten years

SECONDARY OUTCOMES:
Functional Outcome | One to ten years

CONTACTS AND LOCATIONS:
Overall Officials: Joseph E Losee, MD, Principal Investigator — University of Pittsburgh Medical Center; Vijay S Gorantla, MD, PhD, Study Director — University of Pittsburgh Medical Center
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gorantla VS, Brandacher G, Schneeberger S, Zheng XX, Donnenberg AD, Losee JE, Lee WP. Favoring the risk-benefit balance for upper extremity transplantation--the Pittsburgh Protocol. Hand Clin. 2011 Nov;27(4):511-20, ix-x. doi: 10.1016/j.hcl.2011.08.008. PMID 22051391
- [Background] Ravindra KV, Gorantla VS. Development of an upper extremity transplant program. Hand Clin. 2011 Nov;27(4):531-8, x. doi: 10.1016/j.hcl.2011.07.008. Epub 2011 Oct 6. PMID 22051393
- [Background] Lovasik D, Foust DE, Losee JE, Lee WP, Brandacher G, Gorantla VS. Helping hands: caring for the upper extremity transplant patient. Crit Care Nurs Clin North Am. 2011 Sep;23(3):505-17. doi: 10.1016/j.ccell.2011.09.002. PMID 22054824
- [Background] Breidenbach WC, Meister EA, Becker GW, Turker T, Gorantla VS, Hassan K, Kaplan B. A Statistical Comparative Assessment of Face and Hand Transplantation Outcomes to Determine Whether Either Meets the Standard of Care Threshold. Plast Reconstr Surg. 2016 Jan;137(1):214e-222e. doi: 10.1097/PRS.0000000000001893. PMID 26710054
- [Background] Breidenbach WC, Meister EA, Turker T, Becker GW, Gorantla VS, Levin LS. A Methodology for Determining Standard of Care Status for a New Surgical Procedure: Hand Transplantation. Plast Reconstr Surg. 2016 Jan;137(1):367-373. doi: 10.1097/PRS.0000000000001892. PMID 26710038
- [Result] Gorantla VS, Schneeberger S, Moore LR, Donnenberg VS, Zimmerlin L, Lee WP, Donnenberg AD. Development and validation of a procedure to isolate viable bone marrow cells from the vertebrae of cadaveric organ donors for composite organ grafting. Cytotherapy. 2012 Jan;14(1):104-13. doi: 10.3109/14653249.2011.605350. Epub 2011 Sep 12. PMID 21905958
- [Result] Lang RS, Gorantla VS, Esper S, Montoya M, Losee JE, Hilmi IA, Sakai T, Lee WP, Raval JS, Kiss JE, Shores JT, Brandacher G, Planinsic RM. Anesthetic management in upper extremity transplantation: the Pittsburgh experience. Anesth Analg. 2012 Sep;115(3):678-88. doi: 10.1213/ANE.0b013e31825da401. Epub 2012 Jun 28. PMID 22745115
- [Result] Schneeberger S, Gorantla VS, Brandacher G, Zeevi A, Demetris AJ, Lunz JG, Metes DM, Donnenberg AD, Shores JT, Dimartini AF, Kiss JE, Imbriglia JE, Azari K, Goitz RJ, Manders EK, Nguyen VT, Cooney DS, Wachtman GS, Keith JD, Fletcher DR, Macedo C, Planinsic R, Losee JE, Shapiro R, Starzl TE, Lee WP. Upper-extremity transplantation using a cell-based protocol to minimize immunosuppression. Ann Surg. 2013 Feb;257(2):345-51. doi: 10.1097/SLA.0b013e31826d90bb. PMID 23001085